CLINICAL TRIAL: NCT06467929
Title: Prospective Collection of Endoscopic and Histopathologic Data from Endoscopic Procedures Performed in UZ Gent
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: ONZ-2022-0177
Record Dates: First submitted 2024-06-14; First posted 2024-06-21 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Endoscopy
Keywords: endoscopy; histopathology; database

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This is an observational study in which images (photos and/or videos of lesions found during endoscopy) will be collected and the associated data about these lesions (size, location in the body, outcome of histology, if resected and examined).

The images will be taken while performing a diagnostic or therapeutic endoscopy. This footage can be recorded in different light modalities, and various lesions can be removed during one procedure. It is of importance that the images are recorded in the best possible image quality.

The images can be either endoscopic images or endoscopic images combined with room view (this means that the endoscopic room can be filmed, for example, to visualize the endoscopist and thus show techniques of the procedure, without the patient being identified). The GDPR regulations will be respected at all times during the video recordings.

The purpose of this registry is to create a database with images in the form of photos and video clips, histopathological data, demographic data of patients and data about the endoscopic procedure. The recording of this data is standard with every endoscopic procedure that patients undergo at UZ Gent.

The data will be used for the following purposes: linking procedural outcomes with procedural data and patient data to improve endoscopic technique and to guarantee quality in our endoscopic unit. In this way the investigators will also be able to identify trends and link adverse events back to the patient data with the aim of informing the patient. In addition, as a university center, the investigators can train doctors in training with this educational material. The footage can be shared via online and/or live presentations that are only accessible to/by healthcare workers and without the patient being identifiable. Such material and its dissemination is essential to improve (the safety of) techniques (such as those of today), to share knowledge about techniques, and in this way to train the next generation of doctors and nurses.

DETAILED DESCRIPTION:
Background Endoscopy and more specifically polypectomy during endoscopy is well established as an effective way of reducing cancer mortality. The majority of lesions detected and removed at colonoscopy are adenomas <10mm in size without advanced histology. These lesions have a low risk of progression to malignancy and are relatively easily removed by standard snare polypectomy with low complication rates. Polyps that are sessile or flat and greater than 20mm in size are found in approximately 1% of all colonoscopies and are more difficult to manage. These lesions, known as large sessile lesions (LSL), have a high rate of advanced histology. Traditionally they have been managed by referral for open or laparoscopic surgery, which is definitive, but invasive, costly, and associated with a significant mortality risk in patients with advanced age or comorbidities. Endoscopic Mucosal Resection (EMR) has emerged in recent years as an alternative to surgery that is now becoming the standard of care. It is an outpatient procedure which is effective, safe and less costly than surgery when delivered at a tertiary referral centre.

Prospective studies have been successful in addressing several aspects of the resection of LSL, producing robust information on the efficacy of the procedure, recurrence rates, bleeding complications and mortality and costs when compared to surgery. Assessment and management strategies for bleeding and deep mural injury or perforation have been derived from analysis of the data. Snare tip soft coagulation of the resection margin post-EMR has been shown to reduce recurrence in a randomised controlled trial.

There remain a number of unanswered questions regarding the endoscopic resection of large lesions and a new study incorporating a greater number of endoscopy units around the world will allow these to be addressed as well as answer questions on the clinical effectiveness of the technique. Enhancing the prediction of submucosal invasive cancer, advanced lesion classification, validation of the assessment of deep injury, treatment of lesion margins post resection to reduce recurrence, prevention and prophylaxis of bleeding, and subtype analyses of the different histological groups of colonic lesions will be examined.

In addition, other techniques such as endoscopic submucosal dissection (ESD) and full thickness resection (FTR) have emerged in recent years and require assessment of their performance versus endoscopic mucosal resection in prospective observational studies.

The same techniques (EMR and ESD) are used to resect lesions in the upper gastrointestinal tract (oesophagus, stomach, and small intestine) and the same prospective observations are necessary to assess effectiveness of these techniques and outcomes to improve future upper gastrointestinal endoscopy.

Trial objectives This monocenter trial aims to prospectively collect video material, images and data of diagnostic and therapeutic endoscopic procedures and the data of the follow up. The imaging during the endoscopy can be done in white light, narrow-band imaging (NBI), blue-light imaging (BLI), I-scan, linked-color imaging or any other available image enhancement technique, including dye-enhancement with indigo carmine or methylene blue.

The aim of this study is to collect these data prospectively in het UZ Gent. The collected videos, images and data will be used for educational (education and/or training of fellows, publications and postgraduate education) or scientific (discussion amongst peers, scientific meetings and presentations and medical research) purposes by all participating sites.

Endpoint Creation of a large digital database of prospectively collected images, videos and data of endoscopic procedures using any type of imaging technique (e.g., white light endoscopy, video chromoendoscopy, …) and with consecutive resection of lesions providing a corresponding histology report.

ELIGIBILITY:
Inclusion Criteria:

* Age => 18 years
* Referral for a surveillance, diagnostic or therapeutic endoscopy
* Digital video material of the endoscopic procedure
* Digital images of the endoscopic procedure
* Videos and/or images can be made in white light or any virtual of dye-based enhancement technique
* Endoscopic procedures performed after IRB approval for this study
* Material collected in adult patients of all sex or race, including pregnant women

Exclusion Criteria:

* Age < 18 years
* Any contraindication to undergo an endoscopic procedure
* Patient did not sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred for a surveillance, diagnostic or therapeutic endoscopy
Sampling Method: Probability Sample
Enrollment: 510 (Estimated)
Dates: Start 2022-12-22 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Digital Database of Prospectively collected images, videos and data of endoscopic procedures | 01/11/2022 - 30/10/2025
  Creation of a large digital database of prospectively collected images, videos and data of endoscopic procedures using any type of imaging technique (e.g., white light endoscopy, video chromoendoscopy, …) and with consecutive resection of lesions providing a corresponding histology report.

CONTACTS AND LOCATIONS:
Overall Officials: David Tate, Doctor, Principal Investigator — UZ Gent
Locations (1):
- University Hospital Ghent, Ghent, East Flanders, Belgium